CLINICAL TRIAL: NCT00426842
Title: A Dose Response Trial Using 5 and 10 mg. of Midodrine Hydrochloride to Treat Orthostatic Hypotension in Persons With SCI
Brief Title: A Dose Response Trial Using 5 and 10 Mg of Midodrine Hydrochloride
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Scientist, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00893; VA Project #5481-06-051 (Other: JJPVAMC IRB)
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Orthostatic Hypotension; Spinal Cord Injury
Keywords: Blood pressure; Orthostatic hypotension; Spinal Cord Injury; Sympathetic vascular control; Midodrine
MeSH Terms: conditions — Hypotension, Orthostatic; Spinal Cord Injuries | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Blood pressure response during HUT following administration of Midodrine Hydrochloride compared with no drug.
  Interventions: Drug: Midodrine Hydrochloride

INTERVENTIONS:
Drug: Midodrine Hydrochloride — Alpha1-agonist, exerts its actions via activation of the alpha-adrenergic receptors of the arteriolar and venous vasculature, producing an increase in vascular tone and elevation of blood pressure.

SUMMARY:
With upright postures, there is an immediate redistribution of blood to the dependent circulation; venous return and central venous filling pressure are reduced, resulting in diminution of cardiac output and blood pressure. These hemodynamic alterations stimulate the baroreceptor reflex, which is mediated via the central nervous system to increase peripheral sympathetic vasomotor tone, restoring blood pressure and cardiac output within seconds-to-minutes of the assumption of the upright position. Following SCI, individuals often experience the inability to adjust to postural changes due to disruption of central command of the baroreceptor reflex and reduction in efferent sympathetic neural pathways; consequently, orthostatic hypotension (OH) and symptoms of cerebral hypo-perfusion may ensue. OH is a well-documented phenomenon, which is characterized by a fall in systolic blood pressure of >20 mmHg or diastolic BP of > 10 mmHg within 3 minutes of assumption of an upright posture. As a consequence of OH, many individuals experience symptoms of cerebral hypo-perfusion which include lightheadedness, dizziness, blurry vision, fatigue, nausea, ringing in the ears, cognitive impairment and heart palpitations. Although several investigators have reported increased prevalence of OH during the acute phase of spinal cord injury (SCI), individuals with chronic injury also experience significant falls in blood pressure with seated upright postures. This investigation will examine the effects of an alpha-agonist, midodrine hydrochloride, during head-up tilt on systemic blood pressure, cerebral blood flow and cerebral oxygenation compared to placebo administration in persons with chronic SCI who demonstrate significant orthostatic hypotension during a 24-hour observation study. This is the first study to determine the dose response and efficacy of midodrine to improve orthostatic blood pressure and cerebral blood flow and oxygenation in the SCI population.

DETAILED DESCRIPTION:
In individuals with SCI, blood pressure regulation is altered compared to the non-SCI population and relates to the degree of sympathetic vascular denervation. The inadequate release of norepinephrine with postural change is a primary component of OH and several reports have documented significantly reduced plasma norepinephrine levels in individuals with tetraplegia. Ephedrine sulfate and midodrine hydrochloride, both 1 receptor agonists, are recommended for the treatment of postural hypotension in this population. Although there are case reports documenting improved blood pressure regulation in persons with SCI treated with an 1 receptor agonist, this pharmacological treatment for OH has not been adequately studied in this population. A dose response trial will be used to determine the efficacy of midodrine hydrochloride (5 and 10 mg) compared to no drug at improving systemic blood pressure, cerebral blood flow and oxygenation and at reducing symptomatic hypotension during tilt-table testing in 16 individuals with SCI who manifest significant orthostatic hypotension (total time [minutes] spent with hypotension [ 20% fall in mean arterial pressure from supine laboratory observation] over a 24-hour observation.

Subjects will receive, in an increasing dose manner and on separate days: no drug, 5 and 10 mg of oral midodrine hydrochloride. Oral ingestion of the pill (placebo or midodrine) will be at 30 minutes during the 60 minute supine rest period prior to the head-up tilt maneuver.

A progressive head-up tilt will be utilized in which the table will be adjusted to 15 , 25 , 35 for 5 minutes at each angle and then will be maintained at 45 for 45 minutes or until the subjects experiences symptoms of compromised cerebral blood flow, which include, but are not limited to, light headedness, blurry vision, dizziness and nausea. Throughout each test day, measurements of heart rate, blood pressure, middle cerebral blood flow velocity, and cerebral oxygenation will be obtained. In addition, blood draws will be completed to capture humoral factors responsible for blood pressure regulation.

ELIGIBILITY:
Inclusion Criteria:

* This study will be performed on subjects 18 to 65 years old, with chronic SCI (> 1 year), who are neurologically stable and have demonstrated significant hypotension (total time [proportion 50%] spent with hypotension [systolic BP below 110 mmHg for males and 100 mmHg for females] during a 24-hour observation.

Exclusion Criteria:

* hypertension
* diabetes
* vascular disease
* cardiac disease
* cardiovascular medication
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Wecht, EdD, Principal Investigator — VA Medical Center, Bronx; William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- [Result] Wecht JM, Rosado-Rivera D, Handrakis JP, Radulovic M, Bauman WA. Effects of midodrine hydrochloride on blood pressure and cerebral blood flow during orthostasis in persons with chronic tetraplegia. Arch Phys Med Rehabil. 2010 Sep;91(9):1429-35. doi: 10.1016/j.apmr.2010.06.017. PMID 20801263
- [Result] Wecht JM, Radulovic M, Rosado-Rivera D, Zhang RL, LaFountaine MF, Bauman WA. Orthostatic effects of midodrine versus L-NAME on cerebral blood flow and the renin-angiotensin-aldosterone system in tetraplegia. Arch Phys Med Rehabil. 2011 Nov;92(11):1789-95. doi: 10.1016/j.apmr.2011.03.022. Epub 2011 Jul 16. PMID 21762873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2008-2010
Pre-assignment Details: no subject was excluded from study participate prior to group assignment.
Groups:
- All Participants: All participants underwent a head-up tilt maneuver following no-drug, midodrine 5 mg and midodrine 10 mg, in that order, on seperate study visits. Blood pressure response during HUT following administration of Midodrine Hydrochloride compared with no drug.
Period: Overall Study
Arm/Group | All Participants
Started | 11
Completed | 10
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: brachial artery systolic blood pressure (mmHg)
Time Frame: The difference between the average supine systolic blood pressure and the average systolic blood pressure at 45 degree head-up tilt position.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No-drug | Midodrine 5 mg | Midodrine 10 mg
Number analyzed (Participants) | 11 | 10 | 10
mmHg
  Baseline Blood Pressure | 98 (5) | 97 (5) | 102 (12)
  Head-up Tilt Blood Pressure | 87 (15) | 96 (19) | 109 (22)

ADVERSE EVENTS:
Groups:
- All Participants: Blood pressure response during HUT following administration of Midodrine Hydrochloride compared with no drug.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
A matching placebo tablet was not used and the order of testing was not randomized. The total number of subjects recruited was relatively small and extrapolation to a broader group of individuals with chronic SCI may not be appropriate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No